CLINICAL TRIAL: NCT01850641
Title: A Phase III Study of PA21 With Calcium Carbonate in Hemodialysis Patients With Hyperphosphatemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kissei Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PA1304
Record Dates: First submitted 2013-05-07; First posted 2013-05-09 (Estimated); Results first posted 2018-10-09 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2014-11

CONDITIONS: Hemodialysis; Hyperphosphatemia
Keywords: Hemodialysis; Hyperphosphatemia
MeSH Terms: conditions — Hyperphosphatemia

ARMS (1):
- PA21 (Experimental)
  Interventions: Drug: PA21

INTERVENTIONS:
Drug: PA21

SUMMARY:
The purpose of this study is to investigate the safety and efficacy when administering PA21 with calcium carbonate in hemodialysis patients with hyperphosphatemia for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Receiving stable maintenance hemodialysis 3 times a week
* Dialysis patients with hyperphosphatemia

Exclusion Criteria:

* Patients having history of a pronounced brain / cardiovascular disorder
* Patients having severe gastrointestinal disorders
* Patients having severe hepatic disorders

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2013-04-29 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2013-12-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Multiple Locations, Japan

RESULTS

PARTICIPANT FLOW:
Groups:
- PA21: PA21
Period: Overall Study
Arm/Group | PA21
Started | 35
Completed | 30
Not Completed | 5
Not completed — Physician Decision | 1
Not completed — Decrease in serum phosphorus | 1
Not completed — Decrease in serum calcium | 2
Not completed — Increase in serum ferritin | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set
Arm/Group | PA21
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 35
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Dialysis vintage [Mean (Standard Deviation); unit: months] | 111.1 (87.5)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events
Time Frame: 12 weeks
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | PA21
Number analyzed (Participants) | 35
Participants | 28

2. Secondary Outcome: Serum Phosphorus Concentrations at End of Treatment (Actual Measured Value)
Time Frame: 12 weeks
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | PA21
Number analyzed (Participants) | 35
mg/dL | 4.89 (1.14)

3. Secondary Outcome: Corrected Serum Calcium Concentrations at End of Treatment (Actual Measured Value)
Time Frame: 12 weeks
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | PA21
Number analyzed (Participants) | 35
mg/dL | 9.52 (0.88)

4. Secondary Outcome: Serum Intact-PTH Concentrations at End of Treatment (Actual Measured Value)
Time Frame: 12 weeks
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | PA21
Number analyzed (Participants) | 35
pg/mL | 177.9 (146.4)

5. Secondary Outcome: Serum Ferritin Concentrations at End of Treatment (Actual Measured Value)
Time Frame: 12 weeks
Population: Safety Set
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | PA21
Number analyzed (Participants) | 35
ng/mL | 73.8 [38.2 to 183.0]

6. Secondary Outcome: TSAT at End of Treatment (Actual Measured Value)
Time Frame: 12 weeks
Population: Safety Set
Measure: Mean (Standard Deviation); unit: percentage of TSAT
Arm/Group | PA21
Number analyzed (Participants) | 35
percentage of TSAT | 27.72 (8.27)

7. Secondary Outcome: Hb Concentrations at End of Treatment (Actual Measured Value)
Time Frame: 12 weeks
Population: Safety Set
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | PA21
Number analyzed (Participants) | 35
g/dL | 11.22 (1.19)

8. Secondary Outcome: Constipation Condition
Time Frame: 12 weeks
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | PA21
Number analyzed (Participants) | 35
Participants
  Week 0: Not at all bothersome | 15
  Week 0: Bothers me very little | 14
  Week 0: Somewhat bothersome | 2
  Week 0: Bothers me quite a lot | 4
  Week 0: Could not tolerate | 0
  End of treatment: Not at all bothersome | 26
  End of treatment: Bothers me very little | 5
  End of treatment: Somewhat bothersome | 2
  End of treatment: Bothers me quite a lot | 2
  End of treatment: Could not tolerate | 0

9. Secondary Outcome: Satisfaction With Bowel Movement
Time Frame: 12 weeks
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | PA21
Number analyzed (Participants) | 35
Participants
  Week 0: Very much satisfied/Satisfied | 21
  Week 0: Can say neither | 8
  Week 0: Very much dissatisfied/Dissatisfied | 6
  End of treatment: Very much satisfied/Satisfied | 28
  End of treatment: Can say neither | 5
  End of treatment: Very much dissatisfied/Dissatisfied | 2

ADVERSE EVENTS:
Arm/Group | PA21
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 1/35
Other Adverse Events (participants affected / at risk) | 23/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PA21 (N=35)
Hepatitis acute (Hepatobiliary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PA21 (N=35)
Nasopharyngitis (Infections and infestations) | 10
Diarrhoea (Gastrointestinal disorders) | 14
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Wound (Injury, poisoning and procedural complications) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No